CLINICAL TRIAL: NCT04513561
Title: Evaluation of the Impact of Lock Down and End of Lock Down on the Management of Patients With Inflammatory and Dysimmune Diseases Followed in the Context of IMMINeNT FHU (Rheumatology, Dermatology, Internal Medicine, Pneumology, Gastroenterology, Neurology).
Brief Title: Evaluation of the Impact of Lock Down and End of Lock Down on the Management of Patients With Inflammatory and Dysimmune Diseases Followed in the Context of IMMINeNT FHU and COVID-19
Acronym: CONFIMID
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_51; 2020_A01596_33 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2020-10

CONDITIONS: Inflammatory Disease; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This questionnaire is distributed via a mailing list (e-mail) of patients treated within the framework of the FHU for pathologies including chronic inflammatory bowel diseases or IBD (Crohn's disease and ulcerative colitis), inflammatory rheumatic diseases (such as rheumatoid arthritis and ankylosing spondylitis), but also asthma, psoriasis, atopic dermatitis as well as systemic autoimmune (such as scleroderma, lupus, angioedema) and neurological (multiple sclerosis) diseases.

A two-step analysis will be conducted: impact of lock down(March 17, 2020 - May 11, 2020) and a 2-month assessment of end of lock down (from May 11, 2020) on issues addressing: overall impact, impact on the disease, treatment and follow-up, and access to information related to the epidemic during these periods.

ELIGIBILITY:
Inclusion Criteria:

patient followed for :

* Chronic inflammatory bowel disease or IBD (Crohn's disease and ulcerative colitis),
* Inflammatory rheumatism (rheumatoid arthritis and spondylitis)
* Multiple Sclerosis
* Asthma
* Psoriasis
* Atopic Dermatitis
* Systemic autoimmune diseases (scleroderma and lupus)

Exclusion Criteria:

* Minor patient
* Patient cannot read or write
* Patient without computer equipment
* Patient with no internet access
* Patient not having filled in his e-mail in his file
* Patient does not wish to be contacted by email

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients Inflammatory and Dysimmune Diseases Followed in the Context of IMMINeNT FHU IMMINeNT FHU (Rheumatology, Dermatology, Internal Medicine, Pneumology, Gastroenterology, Neurology).
Sampling Method: Non-Probability Sample
Enrollment: 921 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
The answer will be considered positive if the patient answers "totally agree", or "agree", or "slightly agree", or "neither agree nor disagree". | At 2 months
  The answer to question 13 of the lock down questionnaire: "Do you feel that you have been less well followed by your medical specialist compared to the pre-lock down period? "

SECONDARY OUTCOMES:
Proportion of patients (in percentage and numbers) whose response is considered positive if the patient answered "Slightly agree", "Agree" or "Totally agree" to question 9 of the lock down questionnaire | At 2 months
Proportion of patients (in percentage and numbers) whose response is considered positive if the patient answered "yes" to question 34 of the lock down questionnaire | At 2 months
Proportion of patients (in percentage and numbers) whose response is considered positive if the patient answered "Slightly agree" or "Agree" or "Strongly agree" to question 38 of the lock down questionnaire | At 2 months
Proportion of patients (in percentages and numbers) whose response will be considered positive to questions 13 and 14 of the lock down questionnaire and comparison between the different specialities filled in in question 3. | At 2 months
  Proportion of patients (in percentages and numbers) whose response will be considered positive if the patient answers "totally agree", or "agree", or "slightly agree", or "neither agree nor disagree" to questions 13 and 14 of the lock down questionnaire and comparison between the different specialities filled in in question 3.
Proportion of patients (in percent and numbers) whose response will be considered positive to questions 9, 13, 14, 38 or "Yes" to question 34 of the end of lock down and lock down Evaluation Questionnaire. | At 2 months
  Proportion of patients (in percent and numbers) whose response will be considered positive if the patient answers "Slightly agree", "Agree" or "Strongly agree" to questions 9, 13, 14, 38 or "Yes" to question 34 of the end of lock down and lock down Evaluation Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric DEZOTEUX, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France